CLINICAL TRIAL: NCT04155567
Title: A Single Center, Open-Label, Phase 1 Study to Evaluate the Pharmacokinetics, Safety and Tolerability of TAK-123 After Intravenous Infusion in Japanese Healthy Adult Male Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics (PK), Safety and Tolerability of TAK-123 After Intravenous Infusion in Japanese Healthy Adult Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-123-1001; U1111-1237-4920 (Other: WHO); JapicCTI-195027 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2019-11-06; First posted 2019-11-07 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- TAK-123 (Experimental): TAK-123 as 3.75 gram per square meter (g/m^2) of sodium phenylacetate and 3.75 g/m^2 of sodium benzoate, intravenous administration over 90 minutes, followed by TAK-123 as 3.75 g/m^2 of sodium phenylacetate and 3.75 g/m^2 of sodium benzoate, intravenous administration over 24 hours.
  Interventions: Drug: TAK-123

INTERVENTIONS:
Drug: TAK-123 — TAK-123 infusion

SUMMARY:
The purpose of this study is to evaluate the PK, safety and tolerability of phenylacetate and benzoate after intravenous administration of TAK-123 in Japanese healthy adult male participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-123. TAK-123 is being tested in Japanese healthy adult men. This study will look at the PK, safety and tolerability of phenylacetate and benzoates of people who administered TAK-123.

The study will enroll approximately 10 participants. All participants will be administered TAK-123 intravenously at the dose level of 3.75 g/m^2 of sodium phenylacetate and 3.75 g/m^2 of sodium benzoate.

- TAK-123 as 3.75 g/m^2 of sodium phenylacetate and 3.75 g/m^2 of sodium benzoate

This single-center trial will be conducted in Japan. The overall time to participate in this study is approximately 8 days. Participants will make multiple visits to the clinic and be hospitalized for four days.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is capable of understanding and complying with protocol requirements in the opinion of the investigator or sub-investigator.
2. The participant signs and dates a written informed consent form prior to the initiation of any study procedures.
3. The participant is a Japanese healthy adult male.
4. The participant is aged 20 to 45 years inclusive at the time of informed consent.
5. The participant weighs at least 50.0 kilogram (kg), and has a body mass index (BMI) between 18.5 and 25.0 kilogram per square meter (kg/m^2), inclusive, at Screening.
6. The participant is sterile, vasectomized or agrees to use an appropriate method of contraception throughout the treatment period.

Exclusion Criteria:

1. The participant has received any investigational drugs within 90 days before screening for this study (including the cases that at least 5 times the elimination half-lives of any investigational drugs have not yet passed).
2. The participant previously received TAK-123, its ingredients, or related compound before participation in this study except for the cases where benzoic acid is ingested as a food additive.
3. The participant is an employee of the study site, or immediate family member, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (example, spouse, parent, child, sibling) or who may be forced to provide consent.
4. The participants have previous or current history of diseases that may affect the participation in this study or study results, including uncontrolled, clinically relevant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, endocrine, hematologic, immune, skin disease or psychiatric disorder.
5. The participant has a history of multiple episodes or severe allergies (example, food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerance to prescription drugs, over-the-counter (OTC) drugs or foods.
6. The participant has had an anaphylactic reaction to active ingredients or additives of TAK-123, ondansetron or additives of ondansetron, or salicylic acid associated with the intravenous administration of TAK-123.
7. The participant has a positive urine drug test at the time of screening.
8. The participant has a history of drug abuse (defined as any illicit drug use) or has a history of alcohol dependence within 2 years before the start of screening or is unwilling to agree to abstain from alcohol and drugs throughout the study.
9. The participant consumes 6 or more servings of caffeinated beverages (containing about 720 milligram [mg] of caffeine or more) such as coffee, tea, cola, or energy drinks per day.
10. The participant is a smoker who smoked cigarettes or used nicotine-containing products (such as nicotine patch) within 6 months before the study drug administration.
11. The participant has a history of cancer.
12. The participant has a positive test result for any of the following at the time of screening: hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody/antigen, serological test for syphilis.
13. The participant has poor peripheral venous access.
14. The participant has undergone whole blood collection of at least 200 milliliter (mL) within 4 weeks (28 days) or at least 400 mL within 12 weeks (84 days) prior to the start of the study drug administration.
15. The participant has undergone whole blood collection of at least 800 mL in total within 52 weeks (364 days) prior to the start of the study drug administration.
16. The participant has undergone blood component collection within 2 weeks (14 days) prior to the start of the study drug administration.
17. The participant has any clinically relevant abnormality in vital signs or 12-lead electrocardiogram (ECG) at screening or predose of Day 1.
18. The participant has abnormal laboratory test values at screening indicating clinically relevant underlying disease, or showing alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5 × upper limit of normal (ULN).
19. The participant has been on an abnormal diet (example, excessive drinking and eating or starvation condition) during the four weeks (28 days) prior to the start of the study drug administration in the opinion of the investigator or sub-investigator.
20. The participant who used or plans to use excluded concomitant medications, supplements, or dietary products during the predefined period in this study.
21. The participant is unlikely to comply with the protocol requirements or is unsuitable as a participant of this study for any other reason in the opinion of the investigator or sub-investigator.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Sekino Clinical Pharmacology Clinic, Toshima-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be reidentified (due to the limited number of study participants/study sites).

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/5f6b603c4db2bf003ab4a363

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 13 November 2019 to 06 December 2019.
Pre-assignment Details: Healthy Japanese male participants were enrolled in the study to receive TAK-123 3.75 gram per square meter (g/m^2) sodium phenylacetate (NaPA) and 3.75 g/m^2 sodium benzoate (NaBZ), as loading dose followed by an equivalent maintenance dose.
Groups:
- TAK-123 3.75 g/m^2 NaPA and NaBZ: TAK-123 3.75 g/m^2 NaPA and TAK-123 3.75 g/m^2 NaBZ as loading dose, infusion, intravenously over 90 minutes, followed by TAK-123 3.75 g/m^2 NaPA and TAK-123 3.75 g/m^2 NaBZ maintenance dose, infusion, intravenously over 24 hours on Day 1.
Period: Overall Study
Arm/Group | TAK-123 3.75 g/m^2 NaPA and NaBZ
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who received at least one dose of TAK-123.
Arm/Group | TAK-123 3.75 g/m^2 NaPA and NaBZ
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (5.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 10
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 173.7 (5.03)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 65.68 (6.994)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m˄2)] | 21.74 (1.532)
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 8
  Former Smoker | 2
Alcohol Classification [Count of Participants; unit: Participants]
  Drank A Few Times Per Month | 5
  Never Drank | 5
Caffeine Classification [Count of Participants; unit: Participants]
  Had Caffeine Consumption | 1
  Had No Caffeine Consumption | 9

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Time Frame: Day 1 up to Day 8
Population: The safety analysis set was defined as all participants who received at least one dose of TAK-123.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-123 3.75 g/m^2 NaPA and NaBZ
Number analyzed (Participants) | 10
Participants | 6

2. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Phenylacetate, Benzoate, and Their Metabolites (Phenylacetylglutamine and Hippurate)
Time Frame: Day 1: pre-infusion and 0.25, 0.75, 1.5, 2.5, 4.5, 6.5, 8.5, 10.5, 12.5, 16.5, 25.5, 26, 26.5, 27, 27.5, 28, 28.5, 29.5, 30.5, 32.5 and 48 hours post-infusion
Population: The pharmacokinetics (PK) analysis set was defined as all participants who received at least one dose of TAK-123 and provided sufficient PK measurements available to estimate at least one estimable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | TAK-123 3.75 g/m^2 NaPA and NaBZ
Number analyzed (Participants) | 10
microgram per milliliter (mcg/mL)
  Phenylacetate | 300.7 (5.2)
  Benzoate | 233.2 (6.9)
  Phenylacetylglutamine | 69.77 (19.8)
  Hippurate | 54.13 (18.0)

3. Primary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Phenylacetate, Benzoate, and Their Metabolites (Phenylacetylglutamine and Hippurate)
Time Frame: as for outcome 2
Population: The PK analysis set was defined as all participants who received at least one dose of TAK-123 and provided sufficient PK measurements available to estimate at least one estimable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram per milliliter (h*mcg/mL)
Arm/Group | TAK-123 3.75 g/m^2 NaPA and NaBZ
Number analyzed (Participants) | 10
hour*microgram per milliliter (h*mcg/mL)
  Phenylacetate | 3931 (22.6)
  Benzoate | 752.6 (16.7)
  Phenylacetylglutamine | 1135 (16.2)
  Hippurate | 413.5 (22.2)

4. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Phenylacetate, Benzoate, and Their Metabolites (Phenylacetylglutamine and Hippurate)
Time Frame: as for outcome 2
Population: The PK analysis set was defined as all participants who received at least one dose of TAK-123 and provided sufficient PK measurements available to estimate at least one estimable PK parameter. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given categories.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | TAK-123 3.75 g/m^2 NaPA and NaBZ
Number analyzed (Participants) | 10
h*mcg/mL
  Phenylacetate | 3932 (22.6)
  Benzoate: number analyzed (Participants) | 0
  Phenylacetylglutamine | 1140 (16.4)
  Hippurate: number analyzed (Participants) | 9
  Hippurate | 427.3 (21.2)

ADVERSE EVENTS:
Time Frame: TEAEs are adverse events (AEs) that started after first dose of study drug up to Day 8
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-123 3.75 g/m^2 NaPA and NaBZ
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-123 3.75 g/m^2 NaPA and NaBZ (N=10)
Sinus tachycardia (Cardiac disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT04155567/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT04155567/SAP_001.pdf